CLINICAL TRIAL: NCT04139954
Title: Observational Registry (BioSTaR) Including Demographic and Clinical Data of Patients Diagnosed With Rheumatoid Arthritis and Spondyloarthritis Using a Biological and Targeted Synthetic Disease Modifying Drug
Brief Title: Observational Registry of Patients With Rheumatoid Arthritis /Spondyloarthritis Using Biological or Targeted Synthetic DMARDs
Acronym: BioSTaR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turkish League Against Rheumatism (Other)
Responsible Party: Principal Investigator, Fatma Gül Yurdakul, Clinical Associate Professor (Fatma Gül Yurdakul), Turkish League Against Rheumatism
Other Study IDs: TRASD
Record Dates: First submitted 2019-09-01; First posted 2019-10-25 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis and Spondyloarthritis: Patients using Biological or Targeted Synthetic DMARDs
  Interventions: Other: There is no intervention in the study

INTERVENTIONS:
Other: There is no intervention in the study — There is no intervention in the study

SUMMARY:
In this study, investigators aimed to observe the examination findings, laboratory findings and drugs used in routine polyclinic controls of the participants using biological and targeted synthetic disease-modifying antirheumatic drug (DMARD) and the doses and side effects of these drugs. The aim of this registry is to evaluate the real-life data of participants receiving these medications. Analysis of treatment follow-up, drug changes, causes of change, treatment-related paradoxic / immune reactions, compliance with adult vaccination programs, nutritional profiles, presence of metabolic syndrome, fertility status, pregnancy outcomes, and vitamin D levels will be recorded in the outpatient clinic. Rheumatoid Arthritis Impact of Disease, Psoriatic Arthritis Impact of Disease (RAID and PSAID indexes), Work Productivity and Activity Impairment Questionnaire (WPAI), drug compliance, central sensitization and fall risk will be evaluated with verbal evaluation forms performed at policlinic controls in patients with spondyloarthritis and rheumatoid arthritis. It is planned to conduct scientific analyzes and publish on various subjects from the recorded information on this registration system.

Patients using biological and targeted synthetic DMARD treatments are closely monitored and evaluated in many ways due to the risk profiles and various characteristics of the drugs. With this registry system, it is aimed to evaluate the real-life data of the participants using these drugs. Real-life data are very valuable in monitoring the disease and the drugs.

The study is observational and there is no expected risk since no intervention is planned.

DETAILED DESCRIPTION:
In this study, investigators aimed to observe the examination findings, laboratory findings and drugs used in routine polyclinic controls of the participants using biological and targeted synthetic disease-modifying antirheumatic drug (DMARD) and the doses and side effects of these drugs. The aim of this registry is to evaluate the real-life data of participants receiving these medications. Analysis of treatment follow-up, drug changes, causes of change, treatment-related paradoxic / immune reactions, compliance with adult vaccination programs, nutritional profiles, presence of metabolic syndrome, fertility status, pregnancy outcomes, and vitamin D levels will be recorded in the outpatient clinic. Rheumatoid Arthritis Impact of Disease, Psoriatic Arthritis Impact of Disease (RAID and PSAID indexes), Work Productivity and Activity Impairment Questionnaire (WPAI), drug compliance, central sensitization and fall risk will be evaluated with verbal evaluation forms performed at policlinic controls in patients with spondyloarthritis and rheumatoid arthritis. It is planned to conduct scientific analyzes and publish on various subjects from the recorded information on this registration system.

Patients using biological and targeted synthetic DMARD treatments are closely monitored and evaluated in many ways due to the risk profiles and various characteristics of the drugs. With this registry system, it is aimed to evaluate the real-life data of the participants using these drugs. Real-life data are very valuable in monitoring the disease and the drugs.

Planned studies are:

ROMATOID ARTHRITIS CLINICAL DEMOGRAPHIC ASSESSMENT / DISEASE EFFECT / DRUGS

* SPONDYLOARTHRITIS CLINICAL DEMOGRAPHIC EVALUATION / DISEASE EFFECT / DRUGS
* COMORBIDITY IN ROMATOID ARTHRITIS
* COMORBIDITY IN SPONDYLOARTHRITIS
* RE ACTIVITATION AND SAFETY MONITORING IN VIRAL HEPATITIS
* TREATMENT PARADOXIC / IMMUNE REACTIONS (SYSTEMIC AUTOIMMUNE, ARTHRITIS, HEMATOLOGIC, NEUROLOGIC, PULMONARY, OPHTHALMOLOGICAL, INFLAMMATORY BOWEL DISEASE, LIVER, CUTANEOUS, OTHER)
* WORK FORCE LOSS IN AXIAL SPONDYLOARTHRITIS
* WORK FORCE LOSS IN PSORIATIC ARTHRITIS
* WORK FORCE LOSS IN ROMATOID ARTHRITIS
* PREGNANCY / FERTILITY OUTCOMES
* TUBERCULOSIS MONITORING
* DRUG SWITCH ANALYSIS
* THROID DISEASE IN EARLY AND ESTABLISHED ROMATOID ARTHRITIS (AUTOIMMUNE THROIDITIS, MALIGNITY etc)
* TREATMENT COMPLIANCE IN RHEUMATIC DISEASES
* ADULT IMMUNIZATION PROGRAM IN RHEUMATIC DISEASES
* METABOLIC SYNDROME ASSESSMENT
* CARDIOVASCULAR RISK ASSESSMENT
* FALL / FRACTURE AND RELATED VARIABLES IN RHEUMATIC DISEASES
* VITAMIN D STATUS IN RHEUMATIC DISEASES
* CENTRAL SENSITIZATION AND PAIN IN ROMATOID ARTHRITIS AND SPONDYLOARTROPATHIES AND RELATED VARIABLES The study is observational and there is no expected risk since no intervention is planned.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis with rheumatoid arthritis or spondyloarthritis Receiving biological or targeted synthetic DMARD treatment

Exclusion Criteria:

Aged under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients followed in rheumatology and physical medicine and rehabilitation clinics in tertiary hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Disease activity RA | 24 weeks
  DAS 28 score will be calculated (Sensitive and swollen joints, VAS pain score, patient's global assessment and CRP / ESH values will be used for scoring)
Disease activity- SpA1 | 24 weeks
  ASDAS score will be calculated (Sensitive and swollen joints, VAS pain score, patient's global assessment and CRP / ESH values will be used for scoring)
Disease activity-SpA2 | 24 weeks
  BASDAI score will be calculated

OTHER OUTCOMES:
WPAI (Work Productivity and Activity Impairment Questionnaire) | an average of 1 year
  Work Productivity and Activity Impairment Questionnaire:
RAID (Rheumatoid Arthritis Impact of Disease Questionnaire) | an average of 1 year
  Rheumatoid Arthritis Impact of Disease Questionnaire
PSAID (Psoriatic Arthritis Impact of Disease Questionnaire) | an average of 1 year
  Psoriatic Arthritis Impact of Disease Questionnaire
DN-4 (Douleur Neuropathic 4 Questionnaire) questions) | an average of 1 year
  Neuropathic pain questionnaire
Cardiovascular disease risk | 1 year
  HDL and LDL cholesterol (mg/dl) levels from records , hypertension and diabetes history will be evaluated
SF-36 (Short form 36) | an average of 1 year
  Quality of life questionnaire
HAQ (Health assessment questionnaire) | an average of 1 year
  Functional assessment, Questionnaire
ASAS-HI (ASAS Health Index) | an average of 1 year
  ASAS Health Index
Fibromyalgia and central sensitization | an average of 2 year
  Fibromyalgia criteria and central sensitization will be questioned
Demographic characteristics -Age | It will be evaluated at the beginning of the study
  Age, years
Demographic characteristics -Gender | It will be evaluated at the beginning of the study
  female/ male
Demographic characteristics- smoking | It will be evaluated at the beginning of the study
  Amount of smoking (packet-year)
Demographic characteristics- alcohol use | It will be evaluated at the beginning of the study
  How much and how often drink
Demographic characteristics- education | It will be evaluated at the beginning of the study
  Illiterate, literate, years of training
Demographic characteristics- fertility and pregnancy history | It will be evaluated at the beginning of the study
  In her history; pregnancy, abortus, stillbirth, live birth, anomalies number
Demographic characteristics, body mass index (kg/m2) | an average of 2 year
  Height (cm)
Demographic characteristics, body mass index (kg/m2) | an average of 2 year
  Weight (kg)
Demographic characteristics, menopause | It will be evaluated at the beginning of the study
  presence of menopause
Physical examination hand deformities, | It will be evaluated at the beginning of the study
  subluxation, deviation, swan neck, button marrow deformities in hand examination
Physical examination hand deformities, | It will be evaluated at the beginning of the study
  Subcutanea nodules
Lung involvement | an average of 2 year
  Known pulmonary involvement, pulmonary function test and computed tomography results
Neurological involvement | an average of 2 year
  Existing entrapment neuropathy, central involvement will be recorded
Laboratory- Urea | an average of 1 year
  Urea levels from records
Laboratory- creatinine | an average of 1 year
  Creatinine levels from records
Laboratory- liver function tests | an average of 1 year
  Liver function tests from records
Laboratory-vitamin D | an average of 1 year
  Vitamin D levels from records
Laboratory-hemoglobin | an average of 1 year
  hemoglobin levels from records
Laboratory-leukocyte | an average of 1 year
  leukocyte levels from records
Laboratory-platelet | an average of 1 year
  platelet levels from records
Laboratory-Rheumatoid factor (RF) | It will be evaluated at the beginning
  Rheumatoid factor (RF) levels from records
Laboratory-anticyclic citrullinated peptide (Anti CCP) | It will be evaluated at the beginning
  Anti CCP levels from records
Laboratory-Lipid profile | an average of 2 year
  LDL, HDL, Triglycerin, Cholesterol levels from records
Laboratory-hepatitis serology | an average of 2 year
  HBs Ag, Anti HBs, HBc Ag, HBe Ag, Anti HBC levels from records, receiving antiviral treatment for hepatitis, hepatitis reactivation history will be questioned
Laboratory-HIV serology | an average of 2 year
  Anti HIV levels from records
Imaging findings- X Ray | It will be evaluated at the beginning
  Hand wrist and pelvis X ray from records
Imaging findings- magnetic resonance imaging | It will be evaluated at the beginning
  Sacroiliac joint MRI from records
Imaging findings- Ultrasound | It will be evaluated at the beginning
  Hand ultrasound from records
Imaging findings- Bone Mineral density | an average of 2 year
  Bone Mineral density from records
Comorbidity | It will be evaluated at the beginning
  Presence of hypertension, diabetes, autoimmune thyroiditis, metabolic syndrome, coronary artery disease, chronic renal failure,pulmonary dieses, gastric ulcer, anxiety, depression, surgeries, cancer from patient records
Fall risk | It will be evaluated at the beginning
  The number of falls in the last year, the feeling of walking imbalance and the fear of falling and fracture history
Evaluation of tuberculosis | It will be evaluated at the beginning
  PPD / quantiferon result and INH use before drug initiation
Vaccination program | It will be evaluated at the beginning
  Applied hepatitis, tuberculosis, pneumonia, influenza vaccination programme
Drugs | an average of 1 year
  All drugs and doses previously used in relation to rheumatic disease will be questioned. Side effects, autoimmune/ paradoxic reactions and switching of drugs from records will be checked
BASMI | an average of 2 year
  Bath Ankylosing Spondylitis Metrology Index
MASES | an average of 1 year
  Maastricht Ankylosing Spondylitis Enthesitis Score
PASI | an average of 1 year
  The Psoriasis Area Severity Index

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Bodur, Prof Dr, Study Director — Turkish League Against Rheumatism; Şebnem Ataman, Prof Dr, Study Director — Turkish League Against Rheumatism; Fatma G Yurdakul, MD, Principal Investigator — Turkish League Against Rheumatism; Özgür Akgül, AssocProf Dr, Principal Investigator — Turkish League Against Rheumatism; Erhan Çapkın, Prof Dr, Principal Investigator — Turkish League Against Rheumatism; Fatih Çay, AssocProf Dr, Principal Investigator — Turkish League Against Rheumatism; Remzi Çevik, Prof Dr, Principal Investigator — Turkish League Against Rheumatism; Tuncay Duruöz, Prof Dr, Principal Investigator — Turkish League Against Rheumatism; Feride Göğüş, Prof Dr, Principal Investigator — Turkish League Against Rheumatism; Gülcan Gürer, Prof Dr, Principal Investigator — Turkish League Against Rheumatism; Ayhan Kamanlı, Prof Dr, Principal Investigator — Turkish League Against Rheumatism; Meltem Alkan Melikoğlu, Prof Dr, Principal Investigator — Turkish League Against Rheumatism; Aylin Rezvani, AssocProf, Principal Investigator — Turkish League Against Rheumatism; İlhan Sezer, Prof Dr, Principal Investigator — Turkish League Against Rheumatism; İsmihan Sunar, MD, Principal Investigator — Turkish League Against Rheumatism; İlker Yağcı, Prof Dr, Principal Investigator — Turkish League Against Rheumatism
Locations (14):
- Turkey (Türkiye) (14):
  - Ankara Numune Training and Education Hospital, Department of Physical Medicine and Rehabilitation, Ankara
  - Ankara University, Faculty of Medicine, Department of Rheumatology, Ankara
  - Gazi University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Department of Rheumatology, Ankara
  - Akdeniz University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Antalya
  - Antalya Training and Research Hospital Physical Medicine and Rehabilitation Clinic, Antalya
  - Adnan Menderes University, Faculty of Medicine, Department of Rheumatology, Aydin
  - Dicle University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Diyarbakır
  - Istanbul Medipol University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Istanbul
  - Marmara University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Department of Rheumatology, Istanbul
  - Marmara University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Istanbul
  - Celal Bayar University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Manisa
  - Sakarya University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Sakarya
  - Atatürk University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Sivas
  - Karadeniz Technical University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
All of the collected data will be shared with investigators of the study
Supporting Information: Study Protocol, ICF
Time Frame: After the end of the study

REFERENCES:
- [Derived] Bodur H, Yurdakul FG, Ataman S, Cay HF, Gurer G, Capkin E, Sezer I, Duruoz MT, Melikoglu MA, Rezvani A, Yagci I, Gogus F, Kamanli A, Akgul O, Cevik R. Where we are in treat to target era? Predictive factors for remission and drug switching in patients with axial spondyloarthritis: a real-life evidence from BioStaR nationwide registry. Clin Rheumatol. 2022 Jul;41(7):2053-2063. doi: 10.1007/s10067-022-06145-8. Epub 2022 Mar 30. PMID 35353263